CLINICAL TRIAL: NCT06396039
Title: A Phase 4, Multicenter, Single-arm, Open-label Study to Evaluate the Effectiveness and Safety of Oral Ozanimod for Relapsing Multiple Sclerosis (RMS) in Chinese Participants
Brief Title: A Study to Assess the Effectiveness and Safety of Ozanimod in Chinese Adults With Relapsing Multiple Sclerosis
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM047-1096
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — ozanimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Administration of BMS-986374 (Experimental)
  Interventions: Drug: BMS-986374

INTERVENTIONS:
Drug: BMS-986374 — Specified dose on specified days.
  Other Names: Ozanimod

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of ozanimod in Chinese adults with relapsing multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria

* Participants must have Multiple Sclerosis (MS) as diagnosed by the 2017 revision of the McDonald criteria.
* Participants must be exhibiting a relapsing clinical course consistent with Relapsing Multiple Sclerosis (RMS) and history of brain MRI lesions consistent with MS.
* Participants must have an EDSS score between 0 and 5.0 (both inclusive) at baseline.

Exclusion Criteria

* Participants must not have primary progressive MS at screening.
* Participants must not be diagnosed with, or suspected to have neuromyelitis optica spectrum disorder (NMOSD) by clinical symptoms, MRI appearance, and/or supportive serologies according to international consensus criteria.28 A positive test for aquaporin-4 (AQP4) by history or at screening is exclusionary.
* Participants must not have clinically relevant hepatic, neurological, pulmonary, ophthalmological, endocrine, renal, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult or that would put the participant at risk by participating in the study in the opinion of the Investigator.
* Specific cardiac conditions are excluded, including history or presence of:.

  i) Recent (within the past 6 months) occurrence of myocardial infarction, unstable angina, stroke, transient ischemic attack, decompensated heart failure requiring hospitalization, New York Heart Association (NYHA) Class III/IV heart failure, or severe untreated sleep apnea.

ii) Second-degree (Mobitz type II) atrioventricular (AV) block, third-degree AV block, sick sinus syndrome, or sino-atrial block unless participants have a pacemaker in place.

iii) Prolonged corrected QT interval by Fredericia's formula (QTcF; > 450 msec males and > 470 msec females), or participants at additional risk for QT prolongation.

* Participants must not have diabetes mellitus type 1 or uncontrolled diabetes mellitus type 2 with hemoglobin A1c > 9%, or diabetic participants with significant comorbid conditions such as retinopathy or nephropathy.
* Participants must not receive a live vaccine or a live-attenuated vaccine within 4 weeks prior to first dose or planning to receive a live vaccine or a live-attenuated vaccine during the study or within 28 days after discontinuation from study intervention.
* Participants must not have a history of any significant drug allergy (such as anaphylaxis or hepatotoxicity).
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2028-12-29 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Annualized relapse rate (ARR) over 36 months | Up to 3 years

SECONDARY OUTCOMES:
Annualized relapse rate (ARR) over 12 months and 24 months | Up to 2 years
The cumulative number of new or enlarging hyperintense T2-weighted brain MRI lesions at Months 12, 24, and 36 | Up to 3 years
The cumulative number of GdE brain MRI lesions at Months 12, 24, and 36 | Up to 3 years
Proportion of participants who are new or enlarging hyperintense T2 lesion free at Months 12, 24, and 36 | Up to 3 years
Proportion of participants who are GdE lesion-free at Months 12, 24, and 36 | Up to 3 years
Proportion of participants with adverse events (AEs) | Up to 40 months
Proportion of participants with serious adverse events (SAEs) | Up to 40 months
Proportion of participants with AEs leading to discontinuation of study treatment | Up to 3 years
Proportion of participants with laboratory abnormalities | Up to 40 months
Proportion of participants with vital sign abnormalities | Up to 40 months
Proportion of participants with electrocardiogram (ECG) abnormalities | Up to 40 months
Proportion of participants with physical examination abnormalities | Up to 40 months
Proportion of participants with serious or opportunistic infections | Up to 40 months
Proportion of participants with malignancy | Up to 40 months
Proportion of participants with bradycardia and heart condition abnormalities | Up to 40 months
Proportion of participants with pulmonary toxicity | Up to 40 months
Proportion of participants with macular edema | Up to 40 months
Proportion of participants with hepatotoxicity | Up to 40 months
Proportion of participants with posterior reversible encephalopathy syndrome | Up to 40 months
Proportion of participants with progressive multifocal leukoencephalopathy | Up to 40 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (25):
- China (25):
  - Local Institution - 0002, Beijing, Beijing Municipality
  - Local Institution - 0012, Guangzhou, Guangdong
  - Local Institution - 0022, Guangzhou, Guangdong
  - Local Institution - 0008, Shenzhen, Guangdong
  - Local Institution - 0004, Shijiazhuang, Hebei
  - Local Institution - 0006, Harbin, Heilongjiang
  - Local Institution - 0018, Zhengzhou, Henan
  - Local Institution - 0007, Wuhan, Hubei
  - Local Institution - 0003, Nanchang, Jiangxi
  - Local Institution - 0005, Changchun, Jilin
  - Local Institution - 0015, Taiyuan, Shan1xi
  - Local Institution - 0023, Ürümqi, Shan1xi
  - Local Institution - 0016, Shanghai, Shanghai Municipality
  - Local Institution - 0011, Chengdu, Sichuan
  - Local Institution - 0024, Kunming, Yunnan
  - Local Institution - 0019, Hangzhou, Zhejiang
  - Local Institution - 0017, Wenzhou, Zhejiang
  - Local Institution - 0009, Beijing
  - Local Institution - 0025, Fuzhou
  - Local Institution - 0010, Guiyang
  - Local Institution - 0013, Hohhot
  - Local Institution - 0014, Shanghai
  - Local Institution - 0021, Shenyang
  - Local Institution - 0001, Tianjin
  - Local Institution - 0020, Xianyang

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-andresearch/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html